CLINICAL TRIAL: NCT03637400
Title: Short and Long Term Outcomes of Doxycycline Versus Trimethoprim-Sulfamethoxazole for Treatment of Uncomplicated Skin and Soft Tissue Infections
Brief Title: Short and Long Term Outcomes of Doxycycline Versus Trimethoprim-Sulfamethoxazole for Skin and Soft Tissue Infections Treatment
Acronym: TODOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Washington University School of Medicine (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, loren g miller, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30284
Record Dates: First submitted 2018-08-08; First posted 2018-08-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Skin Infection
MeSH Terms: conditions — Cellulitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind trial in which both subjects and study personnel will be masked to the specific treatment arm to which the subject has been assigned and to the results of cultures obtained from the site of infection. The pharmacist will only be unblinded to the liquid formulation, in order to prepare the formulation based upon the subject's weight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trimethoprim/sulfamethoxazole (TMP-SMX) (Experimental): TMP-SMX will be dosed as follows: for adults, 160/800 mg administered as two single strength (SS) over-encapsulated tablets (equivalent to one double strength (DS) tablet) twice daily. As dosages of these medications may be lower in children with lower body weight (<40 kg), we will use weight based liquid medications for children < 40 kg (TMP/SMX dosed based on 8-10 mg/kg of TMP daily, divided into two daily doses) for those children who are under 40 kg in weight. As dosages of these medications are higher in persons with high body weight (>100 kg), we will use TMP/SMX 160/800 mg administered as four single strength (SS) over-encapsulated tablets (equivalent to two double strength (DS) tablet) twice daily.
  Interventions: Drug: TMP-SMX
- Doxycycline (DOXY) (Experimental): DOXY will be dosed as follows: for adults, two 50 mg tabs (100 mg total) given twice daily. As dosages of these medications may be lower in children with lower body weight (<40 kg), we will use weight based liquid medications for children < 40 kg (DOXY 2.2 mg/kg twice daily) for those children who are under 40 kg in weight. The doxycycline dose will remain the same for persons with high body weight (>100 kg) and four additional placebo tabs will be given to subjects > 100 kg randomized to doxycycline.
  Interventions: Drug: DOXY

INTERVENTIONS:
Drug: TMP-SMX — TMP-SMX will be administered over a period of 7 days.
  Other Names: Trimethoprim/sulfamethoxazole
  Arms: Trimethoprim/sulfamethoxazole (TMP-SMX)
Drug: DOXY — DOXY will be administered over a period of 7 days.
  Other Names: Doxycycline
  Arms: Doxycycline (DOXY)

SUMMARY:
The purpose of this study is to compare how well two different antibiotics, doxycycline (DOXY) and trimethoprim/sulfamethoxazole (TMP/SMX), work at curing uncomplicated skin and soft tissue infection (uSSTI) such as 1.Boils (pus in the skin, also known as abscesses and furuncles) or 2. Infections that appear only on the skin surface (called cellulitis and erysipelas) that have pus.

DETAILED DESCRIPTION:
This is a phase IIb multicenter, randomized, double-blind trial in which enrolled subjects with abscess or cellulitis will be treated with either DOXY or TMP-SMX.

The overall objective is to provide a clinically relevant treatment strategy for uSSTI in children and adults in areas where CA-MRSA is prevalent. Out-patient subjects, both children and adults with abscess and/or purulent cellulitis will be enrolled into a randomized, double-blind trial in which enrolled subjects will be treated with either DOXY or TMP-SMX.

Background: Staphylococcus aureus is the most commonly identified cause of skin infections. In the last 15 years, there also has been an large increase in Staphylococcus aureus skin infection attributable to CA-MRSA (Methicillin-resistant Staphylococcus aureus) throughout the United States. However, optimal treatment remains unclear and several commonly used antibiotics such as doxycycline are commonly used but understudied. As resistance among CA-MRSA strains to commonly used antibiotics such as clindamycin continues to increase, there is a need to understand the relative safety and efficacy of alternative treatments, such as doxycycline. This clinical trial will evaluate DOXY and TMP-SMX for the outpatient management of uSSTI in two metropolitan areas, Los Angeles and St. Louis, cities with high prevalence of CA-MRSA. This trial will test important unanswered hypotheses relating to the treatment of CA-MRSA uSSTI and it will advance healthcare providers' ability to successfully manage adults and children with uSSTIs in areas where CA-MRSA is prevalent.

Methods: Out-patient subjects, both children and adults with abscess and/or purulent cellulitis will be enrolled into a randomized, double-blind trial in which enrolled subjects will be treated with either DOXY or TMP-SMX. Using a 1:1 randomized controlled trial of 462 subjects, the investigators aim to 1) compare the cure rate of DOXY to that of TMP-SMX for the treatment of patients throughout the study 2) compare rates of adverse events and of adverse events that are treatment limiting between DOXY and TMP-SMX 3) estimate relapse and recurrence of uSSTI among patients treated with DOXY and of TMP-SMX 4) estimate treatment failure among patients with uSSTI colonized with S. aureus at the anterior nares and oropharynx.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9 years to 85 years
2. Able to complete the informed consent process or, if a minor, a parent or guardian who is able to complete the informed consent process; an assent form also will be completed for children age 9 and older
3. Willing and able to complete the study protocol, study-related activities, and visits
4. Diagnosis of uSSTI, either purulent cellulitis (defined as an inflammation of skin and associated skin structures) or abscess (defined as a circumscribed collection of pus), evidenced by at least 2 of the following localized signs or symptoms on the skin for at least 24 hours:

   1. Erythema
   2. Swelling or induration
   3. Local warmth
   4. Purulent drainage
   5. Tenderness to palpation or pain
5. Pus or drainage from wound that can be sent for clinical culture
6. Able to take oral antibiotic therapy, either in pill or suspension form
7. For women of childbearing potential, the participant agrees to use birth control for the 7 days on the study medication and 7 days after completion of study medication

   Patients who have received prior antibacterial therapy with anti-staphylococcal activity within the prior 14 days:
8. Received prior systemic antibacterial therapy with anti-staphylococcal activity for a skin infection and are not on it currently, and have relapse/recurrence of skin infection.
9. Received prior systemic antibacterial therapy with anti-staphylococcal activity for a skin infection (including those currently on it) without adequate source control of their skin infection and lack of response (i.e., persistence or progression of the lesion) to pre-study antibacterial therapy with on-going evidence of skin infection.
10. Received prior antibiotics with anti-staphylococcal activity for non-skin infections and who developed a skin infection while on these antibiotics or shortly after completing these antibiotics.

Exclusion Criteria:

1. Cellulitis without abscess, drainage, or other culturable exudate.
2. Hospital inpatient
3. Hospitalization within the prior 14 days
4. Residence in a long-term skilled nursing facility
5. Requirement for hospitalization for skin infection or other condition
6. Previous enrollment in this protocol
7. Participation in another clinical trial within the previous 30 days
8. Superficial skin infection only, including

   1. Impetigo
   2. Ecthyma
   3. Folliculitis
   4. Infections that have a high cure rate after surgical incision alone (such as isolated furunculosis) or after topical or local measures
9. Unstable psychiatric or psychological condition rendering the subject unlikely to be cooperative or to complete study requirements
10. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with the adherence or subject compliance with study requirements
11. Systolic blood pressure > 180 mm Hg
12. Systolic blood pressure (SBP) less than an age-specific critical value:

    1. Age 9 to 17 years: < 90 mm Hg
    2. Age ≥ 18 years: < 90 mm Hg
13. Heart rate less than 45 beats per minute (BPM)
14. Heart rate greater than an age-specific-critical value:

    1. Age 9 to 17 years: > 120 BPM
    2. Age ≥ 18 years: > 120 BPM
15. Oral temperature (or equivalent rectal, tympanic membrane, axillary defined in Table 2) less than 35.5° C (95.9° F)
16. Oral temperature (or equivalent rectal, tympanic membrane, axillary defined in Table 2) greater than age-specific critical value:

    1. Age 9 to 17 years: > 38.5° C (101.3° F)
    2. Age ≥ 18 years: > 38.5° C (101.3° F)
17. Documented human or witnessed animal bite in the past 30 days at the site of infection
18. Received prior systemic antibacterial therapy with anti-staphylococcal activity within the prior 14 days who do not meet inclusion criteria 8, 9 and 10.
19. The following concomitant medications: warfarin, phenytoin, methotrexate, dofetilide, methanamine, amiodarone, leucovorin, pyrimethamine, acitretin, atovaquone, atovaquone/proguanil, isotretinoin, or sulfonylureas and systemically administered antibacterial agents with activity against staphylococci
20. Diagnosed or suspected disseminated or severe S. aureus or GAS infection, including lymphangitic spread of skin infection, septicemia, bacteremia, pneumonia, endocarditis, osteomyelitis, septic arthritis, gangrene, necrotizing fasciitis, myositis, or other serious or infections
21. Infection at an anatomical site skin requiring specialized management or specialized antimicrobial therapy, including

    1. Periauricular or orbital infection
    2. Perirectal infection
    3. Suspected deep space infection of the hand or foot
    4. Genital infection
    5. Mastitis
    6. Bursitis
22. Radiographic evidence or suspicion of gas in the tissue or foreign body infection (note: radiography is not required for screening and can be performed at the discretion of the treating physician)
23. Gastrointestinal symptoms such as nausea, vomiting, or diarrhea of a severity that would preclude consumption of oral antibiotics
24. Hypersensitivity or history of allergic reaction to study drug
25. History of G6PD deficiency
26. Pregnant or lactating, or intending to become pregnant within 3 months after screening Women of childbearing potential must have a negative urine or serum pregnancy test result within 1 day prior to initiation of study drug.
27. Severe or morbid obesity with a body mass index (BMI) >45 kg/m2; patients above BMI >45 can be enrolled if their weight is < 100 kg kg/m2.
28. Complicated skin or soft tissue infection, such as

    1. Catheter or catheter site infection within 30 days of placement
    2. Surgical site infection
    3. Known or suspected prosthetic device infection
    4. Suspected Gram-negative or anaerobic pathogen
    5. Unusual exposure history (e.g., underwater injury, fish-tank exposure, heavy soil exposure, etc)
29. History of drug-induced thrombocytopenia and documented megaloblastic anemia due to folate deficiency.
30. Infection at the site of an area of underlying skin disease such as chronic eczema, psoriasis, atopic dermatitis, or chronic venous stasis
31. History of severe underlying immunocompromising condition or immunodeficiency, for example

    1. Chronic renal failure, creatinine clearance <30 ml/min
    2. Renal dialysis within the past 180 days
    3. HIV-positive with either CD4 count <200 or <4% CD4 in the past 180 days or HIV-positive and no documented CD4 count in the past 4 months
    4. Cancer or malignancy with receipt of systemic chemotherapy in the prior 180 days
    5. Organ or bone marrow transplantation (ever), immunosuppressive therapy within the past 180 days, severe liver disease
    6. Other serious underlying disease, as determined by the treating physician or the investigator

Ages: 9 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical cure at Early Clinical Response (ECR) visit | Day 2-3 (48-72 hours)
  Clinical cure is the absence of clinical failure which is defined as occurrence of any one of the following events at ECR:
  * Fever (one or more temperature readings of ≥37.7°C between 48 and 72 hours);
  * Spread of lesion defined as an increase in size (length, width, or area) of the redness, edema, and/or induration such that the size of the lesion is greater than the size at baseline;
  * Administration of rescue antibacterial drug therapy or any non-trial antibacterial drug therapy for the treatment of SSTI prior to the ECR evaluation;
  * Requires an additional unplanned surgical procedure after start of therapy;
  * Death.

SECONDARY OUTCOMES:
Clinical cure at the End of Treatment (EOT) visit | Day 7
  Clinical cure will be defined as complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics is needed
Clinical cure at the One Month Follow-up (OMFU) visit | Day 37
  Clinical cure will be defined as complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics is needed
Adverse events | Day 0-365
  An adverse event (AE) is defined as any unfavorable or undesirable effect (sign, symptom, laboratory abnormality, or condition), regardless of causal relationship to study procedures or participation that occurs in a subject while enrolled in this clinical trial. Any medical condition that is present at the time that the subject is screened should be considered as baseline and not reported as an AE. However, if it deteriorates at any time during the study, it should be recorded as an AE. The occurrence of an AE may come to the attention of study personnel during study visits and interviews of a study recipient presenting for medical care, or upon review by a study monitor.
Adverse events that are treatment limiting | Day 0-365
  An adverse event (AE) is defined as any unfavorable or undesirable effect (sign, symptom, laboratory abnormality, or condition), regardless of causal relationship to study procedures or participation that occurs in a subject while enrolled in this clinical trial. Any medical condition that is present at the time that the subject is screened should be considered as baseline and not reported as an AE. However, if it deteriorates at any time during the study, it should be recorded as an AE. The occurrence of an AE may come to the attention of study personnel during study visits and interviews of a study recipient presenting for medical care, or upon review by a study monitor.
Relapse/recurrent SSTI at One Month Follow-Up (OMFU) | Day 37
  Relapse will be defined as a return of the original infection after initial improvement prior to or at the OMFU visit. Recurrence will be defined as a return of skin infection at the original site, even if considered to be a separate occurrence, after the OMFU visit or a skin infection at a new site of infection.
Relapse/recurrent SSTI at 6 Month Follow-Up (6MFU) | Day 180
  Relapse will be defined as a return of the original infection after initial improvement prior to or at the 6MFU visit. Recurrence will be defined as a return of skin infection at the original site, even if considered to be a separate occurrence, after the 6MFU visit or a skin infection at a new site of infection.
Relapse/recurrent SSTI at 12 Month Follow-Up (12MFU) | Day 365
  Relapse will be defined as a return of the original infection after initial improvement prior to or at the 12MFU visit. Recurrence will be defined as a return of skin infection at the original site, even if considered to be a separate occurrence, after the 12MFU visit or a skin infection at a new site of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Loren G Miller, MD, MPH, Principal Investigator — The Lundquist Institute For Biomedical Innovation at Harbor-UCLA Medical Center; Fritz Stephanie, MD, MSCI, FAAP, FIDSA, FPIDS, Principal Investigator — Washington Univeristy
Locations (3):
- United States (3):
  - Olive View-UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chambers HF. The changing epidemiology of Staphylococcus aureus? Emerg Infect Dis. 2001 Mar-Apr;7(2):178-82. doi: 10.3201/eid0702.010204. PMID 11294701
- [Background] Gorak EJ, Yamada SM, Brown JD. Community-acquired methicillin-resistant Staphylococcus aureus in hospitalized adults and children without known risk factors. Clin Infect Dis. 1999 Oct;29(4):797-800. doi: 10.1086/520437. PMID 10589891
- [Background] Herold BC, Immergluck LC, Maranan MC, Lauderdale DS, Gaskin RE, Boyle-Vavra S, Leitch CD, Daum RS. Community-acquired methicillin-resistant Staphylococcus aureus in children with no identified predisposing risk. JAMA. 1998 Feb 25;279(8):593-8. doi: 10.1001/jama.279.8.593. PMID 9486753
- [Background] Centers for Disease Control and Prevention (CDC). Methicillin-resistant Staphylococcus aureus skin or soft tissue infections in a state prison--Mississippi, 2000. MMWR Morb Mortal Wkly Rep. 2001 Oct 26;50(42):919-22. PMID 11699844
- [Background] Centers for Disease Control and Prevention (CDC). Outbreaks of community-associated methicillin-resistant Staphylococcus aureus skin infections--Los Angeles County, California, 2002-2003. MMWR Morb Mortal Wkly Rep. 2003 Feb 7;52(5):88. PMID 12588006
- [Background] Centers for Disease Control and Prevention (CDC). Methicillin-resistant Staphylococcus aureus infections in correctional facilities---Georgia, California, and Texas, 2001-2003. MMWR Morb Mortal Wkly Rep. 2003 Oct 17;52(41):992-6. PMID 14561958
- [Background] Centers for Disease Control and Prevention (CDC). Methicillin-resistant staphylococcus aureus infections among competitive sports participants--Colorado, Indiana, Pennsylvania, and Los Angeles County, 2000-2003. MMWR Morb Mortal Wkly Rep. 2003 Aug 22;52(33):793-5. PMID 12931079
- [Background] Centers for Disease Control and Prevention (CDC). Methicillin-resistant Staphylococcus aureus skin infections among tattoo recipients--Ohio, Kentucky, and Vermont, 2004-2005. MMWR Morb Mortal Wkly Rep. 2006 Jun 23;55(24):677-9. PMID 16791134
- [Background] Adcock PM, Pastor P, Medley F, Patterson JE, Murphy TV. Methicillin-resistant Staphylococcus aureus in two child care centers. J Infect Dis. 1998 Aug;178(2):577-80. doi: 10.1086/517478. PMID 9697748
- [Background] Ellis MW, Hospenthal DR, Dooley DP, Gray PJ, Murray CK. Natural history of community-acquired methicillin-resistant Staphylococcus aureus colonization and infection in soldiers. Clin Infect Dis. 2004 Oct 1;39(7):971-9. doi: 10.1086/423965. Epub 2004 Sep 2. PMID 15472848